CLINICAL TRIAL: NCT01610362
Title: Human Rabies Immunoglobulin (HRIG)- Dosage Determination and Interference With the Active Immune Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Principal investigator, Queen Saovabha Memorial Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC5504
Record Dates: First submitted 2012-05-29; First posted 2012-06-04 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Rabies
Keywords: rabies; immunoglobulin; dosage
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5-dose IM rabies vaccines, HRIG 20 IU/kg (Active Comparator): Rabies exposed victims, 5-dose IM rabies vaccine, HRIG 20 IU/kg
  Interventions: Biological: Human Rabies Immune Globulin
- 5-dose IM rabies vaccines, HRIG 40 IU/kg (Experimental): Healthy volunteers, 5-dose IM rabies vaccine, HRIG 40 IU/kg
  Interventions: Biological: Human Rabies Immune Globulin

INTERVENTIONS:
Biological: Human Rabies Immune Globulin — HRIG 20 IU/kg and 40 IU/kg would be given once to the volunteers on day 0
  Other Names: Human Rabies Immune Globulin produced by Thai Red Cross

SUMMARY:
Dosage of rabies immune globulin was calculated from the victim's body weight, then the amount of rabies immune globulin would be injected as much as possible to all of the wounds. Increase dosage of rabies immune globulin was needed in situation of multiple severe bite-wounds especially among children whose had lower body weight than adults. Our study would be conducted in order to determine whether the increase dosage of rabies immune globulin would interfere with the protective antibody levels against rabies.

DETAILED DESCRIPTION:
* Controlled trial study.
* All 50 volunteers who had never had rabies immunization would be enrolled and designated into 2 groups.

group 1 : 15 Healthy volunteers age 18 - 60 yr who were attacked by mammals, possible exposed to rabies and had WHO category III exposure, all receive standard post - exposure rabies treatment with 5-dose intramuscular rabies vaccine on day 0,3,7,14,28 and 20 IU/kg of human rabies immune globulin (HRIG).

group 2 : 35 Healthy volunteers age 18 - 60 yr receive 5-dose intramuscular rabies vaccine on day 0,3,7,14,28 and 40 IU/kg of human rabies immune globulin (HRIG).

5 cc - Blood would be drawn from all volunteers before vaccination and on day 14, 28 and 90 for rabies neutralizing antibody titers (RNab).

The GMTs of RNab among both groups would be analyzed and compared.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers age 18-60 years.

Exclusion Criteria:

* received prior rabies immunization
* pregnancy
* immunocompromised conditions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Rabies Neutralizing antibody titers in volunteers who receive HRIG 40 IU/kg | Change from baseline of Rabies Neutralizing Antibody Titers at 3 - month period
  Rabies Neutralizing antibody titers in volunteers who receive HRIG 40 IU/kg would be determined on day 0,14, 28 and 90. Rnab titers above 0.5 IU/ml would be considered as protective levels as WHO recommendation.

SECONDARY OUTCOMES:
Number of participants who have Rabies Neutralizing antibody titers above protective levels. | Number of participants who have Rabies Neutralizing antibody titers above protective levels at 3-month period..
  Number of participants who have Rabies Neutralizing antibody titers above protective levels (> 0.5 IU/mL as recommended by WHO)at 3-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Suda Sibunruang, M.D., Principal Investigator — Queen Saovabha Memorial Institute, Thai Red Cross Society
Locations (1):
- Queen Saovabha Memorial Institute, Thai Red Cross Society, Bangkok, Thailand